CLINICAL TRIAL: NCT05163418
Title: Validation of Plantar Orthoses for Abnormal Plantar Arch Using a New Non-invasive Clinical Imaging System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Cryos Technologies Inc. (Unknown); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD-19-0241_CrA_Valg
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Flat Feet; High Arched Foot
MeSH Terms: conditions — Flatfoot; Talipes Cavus | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flat feet (Experimental): People with flat feet according to foot posture index (validated by clinical assessment)
  Interventions: Device: Foot orthoses for high arches feet
- High arches feet (Experimental): People with high arches feet according to foot posture index (validated by clinical assessment)
  Interventions: Device: Foot orthosis for flat feet
- Normal arches feet (control group) (No Intervention): Control group

INTERVENTIONS:
Device: Foot orthosis for flat feet — Plantar orthotics based on a unique process of footprinting, software design and orthotic printing to create custom 3D printed orthotics.
  Arms: High arches feet
Device: Foot orthoses for high arches feet — Plantar orthotics based on a unique process of footprinting, software design and orthotic printing to create custom 3D printed orthotics.
  Arms: Flat feet

SUMMARY:
The goal of this project is to validate a new non-invasive clinical imaging system to evaluate the efficacy of plantar orthotics and to assess the biomechanical efficiency of plantar orthotics for people with flat or high arch feet. The Cryovizion system should detect changes in participants' posture with an accuracy of 95%, while orthotics should improve the body's postural symmetry index.

ELIGIBILITY:
Inclusion Criteria:

* BMI<30
* No pain
* No musculoskeletal disorders
* No balance disorders
* No pathologies linked to the central nervous system
* No use of drugs affecting the balance

Exclusion Criteria:

* People with foot pathology other than the arch;
* People with diabetes ;
* People with severe obesity ;
* People wearing high heel shoes regularly ;
* People with degenerative disease ;
* People with neuromuscular pathology ;
* People with a circulatory disorder ;
* People who have had major lower body surgery;
* Inability to walk 30 minutes continuously.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edith Martin, PhD, Principal Investigator — TOPMED
Locations (1):
- TOPMED, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flat Feet | High Arches Feet | Normal Arches Feet (Control Group)
Started | 34 | 11 | 20
Completed | 23 | 7 | 20
Not Completed | 11 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Arches Feet (Control Group): Control group. This group only completed the baseline visit, therefore no data is reported for the change from baseline outcome measures.
- Total: Total of all reporting groups
Arm/Group | Flat Feet | High Arches Feet | Normal Arches Feet (Control Group) | Total
Number analyzed (Participants) | 34 | 11 | 20 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 11 | 20 | 65
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 7 | 13 | 46
  Male | 8 | 4 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 34 | 11 | 20 | 65
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 11 | 20 | 65
Body's postural symmetry index [Mean (Standard Deviation); unit: units on a scale] — Body's postural symmetry index(SSIM gray) at baseline. This index is calculated from the full body image based on the Cryovision topographic color imaging system. Index values can range from -1 to 1. 0 indicates no symmetry, 1 indicates perfect symmetry and -1 indicates perfect anti-symmetry.
  units on a scale | 0.348 (0.037) | 0.411 (0.046) | 0.358 (0.039) | 0.361 (0.039)
Asymetry of Flexion/Extension Angle of Lower Body Joints During Gait Without Foot Orthothics [Mean (Standard Deviation); unit: degrees] — Absolute asymmetry values of flexion/extension angle of lower body joints during gait without foot orthotics. The reported values are means of the absolute value of left side flexion/extension joint angle minus right side flexion/extension joint angle. Value=abs(Left joint angle - Right joint angle ). Joint angle values were calculated according to International Society of Biomechanics (ISB) recommandations. Values are reported for hip, knee and ankle asymmetry for gait with shoes but without foot orthotics.
  degrees
    Hip asymmetry | 1.84 (0.94) | 1.90 (1.16) | 1.95 (0.98) | 1.89 (0.98)
    Knee asymmetry | 2.97 (1.27) | 3.14 (1.76) | 3.09 (1.62) | 3.04 (1.47)
    Ankle asymmetry | 2.72 (1.43) | 4.41 (3.06) | 3.77 (3.11) | 3.34 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body's Postural Symmetry Index(SSIM Gray) at 2 Months
Description: Change in body's postural symmetry index(SSIM gray) at 2 months after the beginning of the intervention. This index is calculated from the full body image based on the Cryovision topographic color imaging system. Index values can range from -1 to 1. 0 indicates no symmetry, 1 indicates perfect symmetry and -1 indicates perfect anti-symmetry.
Time Frame: Baseline and 2 months
Population: The normal arches control group only completed the baseline visit, therefore change from baseline outcome measures are not reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: Flat Feet: People with flat feet according to foot posture index 6 (validated by clinical assessment)
- Experimental: High Arches Feet: People with high arches feet according to foot posture index 6 (validated by clinical assessment)
Arm/Group | Experimental: Flat Feet | Experimental: High Arches Feet | Normal Arches Feet (Control Group)
Number analyzed (Participants) | 22 | 7 | 0
score on a scale | -0.031 (0.054) | 0.010 (0.061) |

2. Primary Outcome: Change From Baseline in Body's Postural Symmetry Index(SSIM Gray) at 6 Months
Description: Change in body's postural symmetry index(SSIM gray) at 6 months after the beginning of the intervention. This index is calculated from the full body image based on the Cryovision topographic color imaging system. Index values can range from -1 to 1. 0 indicates no symmetry, 1 indicates perfect symmetry and -1 indicates perfect anti-symmetry.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Flat Feet | Experimental: High Arches Feet | Normal Arches Feet (Control Group)
Number analyzed (Participants) | 22 | 7 | 0
score on a scale | 0.020 (0.070) | -0.016 (0.076) |

3. Primary Outcome: Change From Baseline in Body's Postural Symmetry Index(SSIM Gray) at 12 Months
Description: Change in body's postural symmetry index(SSIM gray) at 12 months after the beginning of the intervention. This index is calculated from the full body image based on the Cryovision topographic color imaging system. Index values can range from -1 to 1. 0 indicates no symmetry, 1 indicates perfect symmetry and -1 indicates perfect anti-symmetry.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Flat Feet | Experimental: High Arches Feet | Normal Arches Feet (Control Group)
Number analyzed (Participants) | 22 | 7 | 0
score on a scale | 0.041 (0.079) | 0.006 (0.057) |

4. Primary Outcome: Change From Baseline in Asymmetry of Flexion/Extension Angle of Lower Body Joints During Gait Without Foot Orthotics at 2 Months
Description: Change from baseline in absolute asymmetry values of flexion/extension angle of lower body joints during gait at 2 months. The reported values are means of the absolute value of left side flexion/extension joint angle minus right side flexion/extension joint angle. Value=abs(Left joint angle - Right joint angle ). Joint angle values were calculated according to International Society of Biomechanics (ISB) recommandations. Values are reported for hip, knee and ankle asymmetry for gait with shoes but without foot orthotics.
Time Frame: Change between directly after 2 months of intervention and baseline values
Population: Participants who completed the overall study.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Experimental: Flat Feet | Experimental: High Arches Feet | Normal Arches Feet (Control Group)
Number analyzed (Participants) | 23 | 7 | 0
degrees
  Hip asymmetry | 0.04 (0.97) | 0.41 (0.33) |
  Knee asymmetry | 0.14 (1.67) | 0.33 (0.81) |
  Ankle asymmetry | 0.20 (1.72) | 0.28 (1.85) |

5. Primary Outcome: Change From Baseline in Asymmetry of Flexion/Extension Angle of Lower Body Joints During Gait Without Foot Orthotics at 6 Months
Description: Change from baseline in absolute asymmetry values of flexion/extension angle of lower body joints during gait at 6 months. The reported values are means of the absolute value of left side flexion/extension joint angle minus right side flexion/extension joint angle. Value=abs(Left joint angle - Right joint angle ). Joint angle values were calculated according to International Society of Biomechanics (ISB) recommandations. Values are reported for hip, knee and ankle asymmetry for gait with shoes but without foot orthotics.
Time Frame: Change between directly after 6 months of intervention and baseline values
Population: Participants who completed the overall study.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Experimental: Flat Feet | Experimental: High Arches Feet | Normal Arches Feet (Control Group)
Number analyzed (Participants) | 23 | 7 | 0
degrees
  Hip asymmetry | 0.09 (0.91) | 0.43 (0.51) |
  Knee asymmetry | 0.27 (1.68) | 0.37 (1.59) |
  Ankle asymmetry | 0.79 (1.81) | 0.18 (1.00) |

6. Primary Outcome: Change From Baseline in Asymmetry of Flexion/Extension Angle of Lower Body Joints During Gait Without Foot Orthotics at 12 Months
Description: Change from baseline in absolute asymmetry values of flexion/extension angle of lower body joints during gait at 12 months. The reported values are means of the absolute value of left side flexion/extension joint angle minus right side flexion/extension joint angle. Value=abs(Left joint angle - Right joint angle ). Joint angle values were calculated according to International Society of Biomechanics (ISB) recommandations. Values are reported for hip, knee and ankle asymmetry for gait with shoes but without foot orthotics.
Time Frame: Change between directly after 12 months of intervention and baseline values
Population: Participants who completed the overall study.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Experimental: Flat Feet | Experimental: High Arches Feet | Normal Arches Feet (Control Group)
Number analyzed (Participants) | 23 | 7 | 0
degrees
  Hip asymmetry | -0.02 (1.10) | 0.28 (0.60) |
  Knee asymmetry | 0.10 (0.94) | 0.47 (1.05) |
  Ankle asymmetry | -0.14 (1.16) | 0.92 (1.87) |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to 12 months visit for the groups with treatment(flat and high arches feet). No follow-up was done with the normal feet group therefore adverse event data was only collected for baseline visit.
Arm/Group | Flat Feet | High Arches Feet | Normal Arches Feet (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/11 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/11 | 0/20
Other Adverse Events (participants affected / at risk) | 4/34 | 4/11 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flat Feet (N=34) | High Arches Feet (N=11) | Normal Arches Feet (Control Group) (N=20)
Foot pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 0 (0) — Foot pain directly associated with the foot orthoses during treatment.

LIMITATIONS AND CAVEATS:
Target number of participants needed to achieve target power was not reached for all groups. Drop outs were not evenly distributed in between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is 1 year from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT05163418/Prot_000.pdf
  • Informed Consent Form (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT05163418/ICF_001.pdf